CLINICAL TRIAL: NCT04277338
Title: SPECT Imaging of Human Epidermal Growth Factor Receptor 2 (HER2) Expression in Breast Cancer Using Technetium-99m-labelled Designed Ankyrin Repeat Proteins HE3-G3 (99mTc-HE3-G3)
Brief Title: Molecular Imaging of HER2 Expression in Breast Cancer Using 99mTc-HE3-G3
Acronym: HE3-G3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Collaborators: Institute of Bioorganic Chemistry, Russian Academy of Sciences (Unknown); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Molecular imaging of HER2
Record Dates: First submitted 2020-02-10; First posted 2020-02-20 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Primary Breast Cancer
Keywords: 99mTc-HE3-G3; Breast Cancer; HER2 expression
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The tested injected doses of 99mTc-HE3-G3 1000 μg (Experimental): At least five (5) evaluable subjects with HER2-positive status and at least five (5) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose. The tested injected dose 1000 μg.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: SPECT
- The tested injected doses of 99mTc-HE3-G3 2000 μg (Experimental): At least five (5) evaluable subjects with HER2-positive status and at least five (5) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose. The tested injected dose 2000 μg.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: SPECT
- The tested injected doses of 99mTc-HE3-G3 3000 μg (Experimental): At least five (5) evaluable subjects with HER2-positive status and at least five (5) subjects with HER2-negative status have to be enrolled in the study for each tested protein dose. The tested injected dose 3000 μg.
  Subjects withdrawn from the study for any reason will be replaced.
  Interventions: Drug: SPECT

INTERVENTIONS:
Drug: SPECT — One single injection of 99mTc-HE3-G3, followed by gamma camera imaging directly postinjection and after 2, 4, 6 and 24 hours.

SUMMARY:
The study should evaluate distribution of 99mTc-HE3-G3 in patients with primary HER2-positive and HER2-negative breast cancer.

The primary objective are:

1. To assess distribution of 99mTc-HE3-G3 in normal tissues and in tumours over time;
2. To evaluate dosimetry of 99mTc-HE3-G3;
3. To obtain initial information concerning safety and tolerability of 99mTc-HE3-G3 after single intravenous injection:

The secondary objective are:

1.To compare the tumour imaging data with the concerning HER2 expression obtained by immunohistochemistry (IHC) or fluorescent in situ hybridisation (FISH) analysis of biopsy samples.

DETAILED DESCRIPTION:
Overall goal of the project: To determine HER2 expression level in primary breast cancer and possibly in axillary lymph node metastases before neoadjuvant trastuzumab therapy.

Phase I. Distribution of 99mTc-HE3-G3 in patients with primary breast cancer. The study should evaluate distribution of 99mTc-HE3-G3 in patients with primary HER2-positive and HER2-negative breast cancer.

The primary objective are:

1. To assess distribution of 99mTc-HE3-G3 in normal tissues and in tumours over time;
2. To evaluate dosimetry of 99mTc-HE3-G3;
3. To obtain initial information concerning safety and tolerability of 99mTc-HE3-G3 after single intravenous injection:

The secondary objective are:

1. To compare the tumour imaging data with the concerning HER2 expression obtained by immunohistochemistry (IHC) or fluorescent in situ hybridisation (FISH) analysis of biopsy samples:

Methodology:

Open-label, exploratory, single centre study. The subjects will receive a single injection of the labelled tracer.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is > 18 years of age
2. Diagnosis of primary breast cancer with possible lymph node metastases
3. Availability of results from HER2 status previously determined on material from the primary tumor, either

   1. HER2-positive, defined as a immunohistochemical test score of 3+ or FISH positive or
   2. HER2-negative, defined as a immunohistochemical test score of 0 or 1+; or else if 2+ then FISH negative
4. Volumetrically quantifiable tumour lesions on CT or MRI, with at least one lesion > 1.0 cm in greatest diameter outside of the liver and kidneys
5. Hematological, liver and renal function test results within the following limits:

   * White blood cell count: > 2.0 x 10^9/L
   * Haemoglobin: > 80 g/L
   * Platelets: > 50.0 x 10^9/L
   * Bilirubin =< 2.0 times Upper Limit of Normal
   * Serum creatinine: Within Normal Limits
6. A negative pregnancy test (serum beta-human chorionic gonadotropin, beta-HCG) at screening for all patients of childbearing potential. Sexually active women of childbearing potential participating in the study must use a medically acceptable form of contraception for at least 30 days after study termination
7. Subject is capable to undergo the diagnostic investigations to be performed in the study
8. Informed consent

Exclusion Criteria:

1. Second, non-breast malignancy
2. Active current autoimmune disease or history of autoimmune disease
3. Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
4. Known HIV positive or chronically active hepatitis B or C
5. Administration of other investigational medicinal product within 30 days of screening
6. Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Gamma camera-based whole-body 99mTc-HE3-G3 uptake value (%) | 6 hours
  Whole-body 99mTc-HE3-G3 uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (%) of the injected dose of the radiopharmaceutical
SPECT-based 99mTc-HE3-G3 uptake value in tumor lesions (counts) | 6 hours
  99mTc-HE3-G3 uptake coinciding with tumor lesions will be assessed using single-photon emission computed tomography and measured in counts
SPECT-based 99mTc-HE3-G3background uptake value (counts) | 6 hours
  Focal uptake of 99mTc-HE3-G3 in the regions without pathological findings will be assessed with SPECT and measured in counts
Tumor-to-background ratio (SPECT) | 6 hours
  The SPECT-based tumor-to-background ratio will be calculated as follows: the value of 99mTc-HE3-G3 uptake coinciding with tumor lesions (counts) will be divided by the value of 99mTc-HE3-G3 uptake coinciding with the regions without pathological findings (counts)

SECONDARY OUTCOMES:
Safety attributable to 99mTc-HE3-G3 injections (physical findings) | 24 hours
  The safety attributable to 99mTc-HE3-G3 injections will be evaluated based on the assessments of physical examination, vital signs, and ECG (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-HE3-G3 injections (laboratory tests) | 24 hours
  The safety attributable to 99mTc-HE3-G3 injections will be evaluated based on the blood and urine laboratory tests (% of cases with abnormal findings relative to baseline)
Safety attributable to 99mTc-HE3-G3 injections (incidence and severity of adverse events) | 24 hours
  The safety attributable to 99mTc-HE3-G3 injections will be evaluated based on the rate of adverse events (%)
Safety attributable to 99mTc-HE3-G3 injections (concomitant medication) | 24 hours
  The safety attributable to 99mTc-HE3-G3 injections will be evaluated based on the rate of administration of concomitant medication (%)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, Principal Investigator — Tomsk NRMC
Locations (1):
- TomskNRMC, Tomsk, Russia

REFERENCES:
- [Derived] Bragina O, Chernov V, Schulga A, Konovalova E, Garbukov E, Vorobyeva A, Orlova A, Tashireva L, Sorensen J, Zelchan R, Medvedeva A, Deyev S, Tolmachev V. Phase I Trial of 99mTc-(HE)3-G3, a DARPin-Based Probe for Imaging of HER2 Expression in Breast Cancer. J Nucl Med. 2022 Apr;63(4):528-535. doi: 10.2967/jnumed.121.262542. Epub 2021 Aug 12. PMID 34385343